CLINICAL TRIAL: NCT04016051
Title: Comparison of Treatment Satisfaction and Treatment Adherence of a Novel Application Form "Dose Sipping Technology" (DST) of Oral Clarithromycin vs. Clarithromycin Syrup in Children Suffering From Acute Otitis Media, Tonsillitis, Pharyngitis, or Acute Bacterial Bronchitis (DoSe iT)
Brief Title: Acceptance of Clarithromycin in a Straw Compared to Syrup in Children With Upper Respiratory Tract Infections
Acronym: DoSe iT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KF-DSTCLA/01
Record Dates: First submitted 2019-06-05; First posted 2019-07-11 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Otitis Media; Tonsillitis; Pharyngitis; Bronchitis
MeSH Terms: conditions — Otitis Media; Tonsillitis; Pharyngitis; Bronchitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clarithromycin DST (Experimental): Participants received oral administration of Clarithromycin DST twice a day:
  * 125.0 mg straw, participants with body weight between 12 and 19 kg (approximate age 2-4 years).
  * 187.5 mg straw, participants with body weight between 20 and 29 kg (approximate age 4-8 years).
  * 250.0 mg straw, participants with body weight between 30 and 40 kg (approximate age 8-12 years).
  For oral intake of DST granules, the lower end of the straw was to be dipped into a glass with a clear, cool or lukewarm, preferably flavored beverage of participant choice. Suitable beverages were lemonade (carbonated or not), clear fruit juices without pulp, tea or water. The beverage was to be sipped smoothly through the straw.
  Interventions: Drug: Clarithromycin DST (125 mg); Drug: Clarithromycin DST (187.5 mg); Drug: Clarithromycin DST (250 mg)
- Clarithromycin Syrup (Active Comparator): Participants received oral administration of Clarithromycin Syrup twice a day:
  * 2.5 ml (125 mg) participants with body weight between 12 and 19 kg (approximate age 2-4 years).
  * 3.75 ml (187.5 mg) participants with body weight between 20 and 29 kg (approximate age 4-8 years).
  * 5 ml (250 mg) participants with body weight between 30 and 40 kg (approximate age 8-12 years).
  Interventions: Drug: Clarithromycin Syrup (125 mg); Drug: Clarithromycin Syrup (187.5 mg); Drug: Clarithromycin Syrup (250 mg)

INTERVENTIONS:
Drug: Clarithromycin DST (125 mg) — Clarithromycin DST (125.0 mg clarithromycin / straw).
  Arms: Clarithromycin DST
Drug: Clarithromycin DST (187.5 mg) — Clarithromycin DST (187.5 mg clarithromycin / straw).
  Arms: Clarithromycin DST
Drug: Clarithromycin DST (250 mg) — Clarithromycin DST (250.0 mg clarithromycin / straw).
  Arms: Clarithromycin DST
Drug: Clarithromycin Syrup (125 mg) — Clarithromycin Syrup 2.5 ml (125 mg).
  Other Names: Klacid Syrup® Forte 250 mg/5mL
  Arms: Clarithromycin Syrup
Drug: Clarithromycin Syrup (187.5 mg) — Clarithromycin Syrup 3.75 ml (187.5 mg).
  Other Names: Klacid Syrup® Forte 250 mg/5mL
  Arms: Clarithromycin Syrup
Drug: Clarithromycin Syrup (250 mg) — Clarithromycin Syrup 5 ml (250 mg).
  Other Names: Klacid Syrup® Forte 250 mg/5mL
  Arms: Clarithromycin Syrup

SUMMARY:
This study was performed in children with upper respiratory tract infections (acute ear infection, infection of the tonsils or throat, or bacterial inflammation of the bronchi) who needed treatment with an antibiotic (clarithromycin). The study investigated a new technology which delivers the antibiotic in a straw (dose sipping technology, DST) in comparison to a marketed syrup.

DETAILED DESCRIPTION:
The study population were children aged 2-12 years (weight 12-40 kg) suffering from upper respiratory tract infections (acute otitis media, tonsillitis, pharyngitis, or acute bacterial bronchitis) and who needed antibiotic treatment. The study compared treatment satisfaction and treatment adherence of oral clarithromycin DST (125 mg, 187.5 mg, or 250 mg twice daily) with the established oral clarithromycin syrup administered via a graduated syringe (Klacid Syrup Forte®, 250 mg/5mL) at the same fixed daily doses.

Fixed doses of 125 mg, 187.5 mg and 250 mg of clarithromycin DST offer the pediatrician the flexibility to treat children of different body weight and age adequately at the recommended daily dose of 15 (12.5-20) mg/kg. All children were treated for 7 to 10 day (14 to 20 doses). Treatment satisfaction by the guardian/caregiver in terms of handling and administration of the clarithromycin DST straw and the comparator clarithromycin syrup, convenience of the administration, acceptance of taste and aftertaste, and treatment satisfaction with respect to future use was evaluated by means of a Parents' Questionnaire once on either Day 3, 4, or 5 and once on either Day 11, 12, 13, or 14. In addition, treatment adherence/willingness of medication intake and the child's health status were assessed. The safety program comprised recording and evaluation of adverse events and countermeasures.

ELIGIBILITY:
Inclusion Criteria:

* Male and female children weighing 12-40 kg.
* Age 2 -12 years.
* Written informed consent (parents).
* Diagnosis of acute otitis media, tonsillitis, pharyngitis, or acute bacterial bronchitis requiring antibiotic treatment.

Exclusion Criteria:

* Participation in another study of investigational products or of devices parallel to, or less than 4 weeks before study entry, or previous participation in this study (for safety reasons).
* Known to or suspected of not being able to comply with the study protocol and the use of clarithromycin.
* Requirement for, or current use of, systemic antibacterial agents not specified in the protocol.
* Necessity of dose reduction due to any concomitant disease.
* Known human immunodeficiency virus (HIV) positive.
* Other inflammatory/infectious diseases of the ear, the upper respiratory tract or the nose and throat.
* History or presence of disease or concomitant medication contraindicating the use of clarithromycin.
* Known or suspected intolerance / hypersensitivity to macrolides.
* Contraindications according to the clarithromycin Summary of Product Characteristics (SmPC).
* Indication for antibiotic treatment for less than 7 days or more than 10 days.
* If known before entry, bacterial isolate resistant to clarithromycin.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 265 (Actual)
Dates: Start 2004-09-22 (Actual); Primary Completion 2004-12-23 (Actual); Study Completion 2004-12-23 (Actual)

PRIMARY OUTCOMES:
Preparation of the medication (during treatment) | Day 3-5
  This was analyzed by a Parents' Questionnaire by means of the question "How was the preparation of the medication?" Parents were asked to respond once on either Day 3, 4, or 5. Possible answers (tick one only) were "very simple", "simple", "complicated" and "very complicated". The best outcome was "very simple", the worst "very complicated". The percentage of responses for each of the possible answers was calculated.
Preparation of the medication (after treatment) | Day 11-14
  This was analyzed by a Parents' Questionnaire by means of the question "How was the preparation of the medication?". Parents were asked to respond once on either Day 11, 12, 13, or 14. Possible answers (tick one only) were "very simple", "simple", "complicated" and "very complicated". The best outcome was "very simple", the worst "very complicated". The percentage of responses for each of the possible answers was calculated.
Dosing accuracy (during treatment) | Day 3-5
  This was analyzed by a Parents' Questionnaire by means of the question "How do you rate giving the right dose?". Parents were asked to respond once on either Day 3, 4, or 5. Possible answers (tick one only) were "very simple", "simple", "difficult" and "very difficult". The best outcome was "very simple", the worst "very difficult". The percentage of responses for each of the possible answers was calculated.
Dosing accuracy (after treatment) | Day 11-14
  This was analyzed by a Parents' Questionnaire by means of the question "How do you rate giving the right dose?" Parents were asked to respond once on either Day 11, 12, 13, or 14. Possible answers (tick one only) were "very simple", "simple", "difficult" and "very difficult". The best outcome was "very simple", the worst "very difficult". The percentage of responses for each of the possible answers was calculated.
Handling of the medication (during treatment) | Day 3-5
  This was analyzed by a Parents' Questionnaire by means of the question "How satisfied are you with the handling of the medication?" Parents were asked to respond once on either Day 3, 4, or 5. Possible answers (tick one only) were "very satisfied", "satisfied", "less satisfied" and "not satisfied". The best outcome was "very satisfied", the worst "not satisfied". The percentage of responses for each of the possible answers was calculated.
Handling of the medication (after treatment) | Day 11-14
  This was analyzed by a Parents' Questionnaire by means of the question "How satisfied are you with the handling of the medication?" Parents were asked to respond once on either Day 11, 12, 13, or 14. Possible answers (tick one only) were "very satisfied", "satisfied", "less satisfied" and "not satisfied". The best outcome was "very satisfied", the worst "not satisfied". The percentage of responses for each of the possible answers was calculated.
Administration of the medication (during treatment) | Day 3-5
  This was analyzed by a Parents' Questionnaire by means of the question "How do you judge the administration of the medication?" Parents were asked to respond once on either Day 3, 4, or 5. Possible answers (tick one only) were "very simple", "simple", "complicated" and "very complicated". The best outcome was "very simple", the worst "very complicated". The percentage of responses for each of the possible answers was calculated.
Administration of the medication (after treatment) | Day 11-14
  This was analyzed by a Parents' Questionnaire by means of the question "How do you judge the administration of the medication?" Parents were asked to respond once on either Day 11, 12, 13, or 14.
  Possible answers (tick one only) were "very simple", "simple", "complicated" and "very complicated". The best outcome was "very simple", the worst "very complicated". The percentage of responses for each of the possible answers was calculated.
Ease to follow the prescribed dosing schedule (during treatment) | Day 3-5
  This was analyzed by a Parents' Questionnaire by means of the question "How easy is it to follow the dosing schedule?" Parents were asked to respond once on either Day 3, 4, or 5. Possible answers (tick one only) were "very simple", "simple", "complicated" and "very complicated". The best outcome was "very simple", the worst "very complicated". The percentage of responses for each of the possible answers was calculated.
Ease to follow the prescribed dosing schedule (after treatment) | Day 11-14
  This was analyzed by a Parents' Questionnaire by means of the question "How easy is it to follow the dosing schedule?" Parents were asked to respond once on either Day 11, 12, 13, or 14. Possible answers (tick one only) were "very simple", "simple", "complicated" and "very complicated". The best outcome was "very simple", the worst "very complicated". The percentage of responses for each of the possible answers was calculated.
Child's feeling about the taste of the medication (during treatment) | Day 3-5
  This was analyzed by a Parents' Questionnaire by means of the question "What does your child feel about the taste of the medication?".
  Possible answers (tick one only) were "very good", "good", "acceptable", "bad", "very bad" and "no comment". The best outcome was "very good", the worst "very bad". The percentage of responses for each of the possible answers was calculated.
Child's feeling about the taste of the medication (after treatment) | Day 11-14
  This was analyzed by a Parents' Questionnaire by means of the question "What does your child feel about the taste of the medication?" Parents were asked to respond once on either Day 11, 12, 13, or 14.
  Possible answers (tick one only) were "very good", "good", "acceptable", "bad", "very bad" and "no comment". The best outcome was "very good", the worst "very bad". The percentage of responses for each of the possible answers was calculated.
Child's feeling about aftertaste of the medication (during treatment) | Day 3-5
  This was analyzed by a Parents' Questionnaire by means of the question "What does your child feel about the aftertaste of the medication?" Parents were asked to respond once on either Day 3, 4, or 5.
  Possible answers (tick one only) were "very good", "good", "acceptable", "bad", "very bad" and "no comment". The best outcome was "very good", the worst "very bad". The percentage of responses for each of the possible answers was calculated.
Child's feeling about the aftertaste of the medication (after treatment) | Day 11-14
  This was analyzed by a Parents' Questionnaire by means of the question "What does your child feel about the aftertaste of the medication?" Parents were asked to respond once on either Day 11, 12, 13, or 14.
  Possible answers (tick one only) were "very good", "good", "acceptable", "bad", "very bad" and "no comment". The best outcome was "very good", the worst "very bad". The percentage of responses for each of the possible answers was calculated.
Optimal administration form | Day 11-14
  This was analyzed by a Parents' Questionnaire by means of the question "Do you think the administration form is optimal for your child?". Parents were asked to respond once on either Day 11, 12, 13, or 14.
  Possible answers (tick one only) were "Yes", "No", and "Do not know". The percentage of responses for each of the possible answers was calculated.
Treatment preference | Day 11-14
  Treatment preference was analyzed by a Parents' Questionnaire by means of the question "Would you or your child prefer this administration form next time?" Parents were asked to respond once on either Day 11, 12, 13, or 14.
  Possible answers (tick one only) were "Yes" and "No". The percentage of responses for each of the possible answers was calculated.
Treatment adherence | Day 11-14
  The child's adherence to the prescribed course of therapy was checked by determining the number of unused straws or the residual volume in the medication bottles, respectively, when unused study medication was returned to the site on Day 11, 12, 13, or 14. A participant was considered to be:
  * Fully treatment adherent: >90 % of prescribed doses taken within the prescribed course of therapy.
  * Partially treatment adherent: 70-90% of prescribed doses taken within the prescribed course of therapy.
  * Non adherent: Omission of 2 or more consecutive doses or <70% of prescribed doses taken within the prescribed course of therapy.
  The percentage of participants in each of the 3 categories was calculated.

SECONDARY OUTCOMES:
Child's Health Status compared to Baseline (during treatment) | Day 3-5
  The participant's overall health status compared to baseline (= acute infection requiring antibiotic treatment) was assessed by the investigator as "cured", "improved", "no changes", or "deteriorated". The clinical assessment was made during a phone interview with the parent/caregiver on either Day 3, 4, or 5. The best outcome was "cured", the worst was "deteriorated". The percentage of participants per outcome category was calculated.
Child's Health Status compared to Baseline (after treatment) | Day 11-14
  The participant's overall health status compared to baseline (= acute infection requiring antibiotic treatment) was assessed by the investigator as "cured", "improved", "no changes", or "deteriorated". The clinical assessment was made once at a site visit on either Day 11, 12, 13. or 14. The best outcome was "cured", the worst was "deteriorated". The percentage of participants per outcome category was calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Grünenthal Study Director, Study Director — Grünenthal GmbH
Locations (20):
- Germany (14):
  - DE11, Balve
  - DE10, Beckum
  - DE09, Hamelin
  - DE08, Hanover
  - DE12, Künzing
  - DE14, München
  - DE05, München
  - DE06, München
  - DE03, München
  - DE02, München
  - DE13, München
  - DE04, Olching
  - DE07, Pullach im Isartal
  - DE01, Unterhaching
- Poland (6):
  - PL03, Koziegłowy
  - PL06, Krakow
  - PL01, LÓDZ
  - PL04, Otwock
  - PL05, Warsaw
  - PL02, Wroclaw

IPD SHARING:
Plan to Share IPD: No